CLINICAL TRIAL: NCT07149454
Title: A Randomized, Double-blind, Controlled, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Intramuscular Injection of Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection in Healthy Participants
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIBP-TAB-01
Record Dates: First submitted 2025-08-03; First posted 2025-09-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Tetanus
Keywords: Tetanus Antitoxin
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (0.2 mg dose group) (Experimental): A single dose was administered to 3 enrolled participants, who were randomized in a 2:1 ratio to receive either the recombinant human anti-tetanus toxin monoclonal antibody injection or placebo. After all participants completed the 14-day safety observation period and were evaluated as safe and tolerable, administration for the next dose group could proceed.
  Interventions: Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection; Drug: Placebo
- Group 2 (2 mg dose group) (Experimental): A single dose was administered to 8 enrolled participants, who were randomized in a 3:1 ratio to receive either the recombinant human anti-tetanus toxin monoclonal antibody injection or placebo. After all participants completed the 14-day safety observation period for the current dose group and were evaluated as safe and tolerable, the trial proceeded to the next dose group.
  Interventions: Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection; Drug: Placebo
- Group 3 (5 mg dose group) (Experimental): A single dose was administered to 15 enrolled participants, who were randomized in a 4:1 ratio to receive either the recombinant human anti-tetanus toxin monoclonal antibody injection or placebo. After all participants completed the 14-day safety observation period for the current dose group and were evaluated as safe and tolerable, the study proceeded to the next cohort.
  Interventions: Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection; Drug: Placebo
- Group 4 (10 mg dose group) (Experimental): A single dose was administered to 27 enrolled participants, who were randomized in a 4:4:1 ratio to receive either:
  the recombinant human anti-tetanus toxin monoclonal antibody injection,
  human tetanus immunoglobulin (HTIG) injection, or
  placebo.
  After all participants completed the 14-day safety observation period for the current dose group and were evaluated as safe and tolerable, the study advanced to the next phase.
  Interventions: Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection; Drug: Human Tetanus Immunoglobulin; Drug: Placebo
- Group 5 (15 mg dose group) (Experimental): A single dose was administered to 15 enrolled participants who were randomized in a 4:1 ratio to receive either the recombinant human anti-tetanus toxin monoclonal antibody injection or placebo.
  As this represented the highest planned dose level, the sponsor and investigators jointly determined whether to continue dose escalation based on the absence of tolerability concerns.
  Interventions: Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection; Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Human Anti-Tetanus Toxin Monoclonal Antibody Injection — intramuscular injection
Drug: Human Tetanus Immunoglobulin — intramuscular injection
  Arms: Group 4 (10 mg dose group)
Drug: Placebo — intramuscular injection

SUMMARY:
A Randomized, Double-blind, Controlled, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Intramuscular Injection of Recombinant Human Anti-tetanus toxin Monoclonal Antibody Injection in Healthy Participants.

DETAILED DESCRIPTION:
The primary objective of the study ： evaluate the safety and tolerability of a single intramuscular injection of recombinant human anti-tetanus toxin monoclonal antibody injection in healthy adult participants. The secondary objectives are:

1. to evaluate the pharmacokinetic (PK) characteristics of a single intramuscular injection of recombinant human anti-tetanus toxin monoclonal antibody injection in healthy adult participants;
2. to evaluate the pharmacodynamic (PD) characteristics of a single intramuscular injection of recombinant human anti-tetanus toxin monoclonal antibody injection in healthy adult participants;
3. to evaluate the immunogenicity of a single intramuscular injection of recombinant human anti-tetanus toxin monoclonal antibody injection in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily agree to participate in the study and sign the informed consent form (ICF);
2. Aged 18-60 years (inclusive) at the time of ICF signing, regardless of gender, with valid legal identification;
3. Body weight ≥45.0 kg for female participants and ≥50.0 kg for male participants, with a body mass index (BMI) between 18.0 and 28.0 kg/m² (inclusive) (BMI = weight [kg]/height [m²]);
4. Female participants of childbearing potential must have no plans for pregnancy or egg donation during the trial and for 6 months after investigational product administration and must voluntarily use at least one effective contraceptive method. Male participants must have no plans for pregnancy or sperm donation during the trial and for 6 months after investigational product administration, and either the male participant or his female partner of childbearing potential must voluntarily use at least one effective contraceptive method.

Exclusion Criteria:

1. Known allergy to the investigational product (including excipients or similar drugs), or documented hypersensitivity to essential materials used in the trial (e.g., skin disinfectants); or history of severe allergic diseases, hypersensitivity to monoclonal antibodies, or allergic constitution deemed by investigators to compromise participant safety;
2. Acute/chronic medical conditions that may significantly affect drug metabolism or safety assessments per investigator judgment;
3. History of autoimmune diseases or immunodeficiency disorders (including HIV-positive screening);
4. Chronic hepatitis B/C (HBsAg or HCV antibody-positive during screening);
5. History/family history of seizures, epilepsy, or neuropsychiatric disorders;
6. Major surgery within 3 months (90 days) prior to dosing, or planned surgery during the trial;
7. Prior tetanus infection or use of passive tetanus immunoglobulins within 6 months (180 days) before dosing;
8. Tetanus-toxoid-containing vaccination (e.g., DTaP, Td, meningococcal conjugate vaccines) within 10 years;
9. Positive tetanus IgG rapid test during screening;
10. Receipt of live/inactivated vaccines within 1 month (30 days) before dosing or planned vaccination during the trial;
11. Systemic corticosteroids/immunosuppressants within 3 months (90 days) (excluding inhaled/topical use);
12. Prescription/OTC/herbal medications within 14 days or <5 half-lives (whichever is longer) prior to dosing, particularly those interfering with the investigational monoclonal antibody's PK/safety (per criterion #11 for exceptions);
13. Participation in other clinical trials involving investigational drugs/devices within 3 months (90 days) or planned concurrent enrollment;
14. Excessive alcohol intake (>14 units/week; 1 unit = 360 mL beer/45 mL 40% liquor/150 mL wine), alcohol use within 48 hours pre-dose, or positive breathalyzer test;
15. Heavy smoking (>10 cigarettes/day or equivalent) within 1 month (30 days);
16. Blood loss/donation >400 mL within 3 months (90 days) or planned donation/transfusion during the trial;
17. Inability to avoid strenuous exercise within 14 days post-dosing;
18. Substance abuse history or positive drug screening;
19. Positive syphilis antibody test during screening;
20. Clinically significant abnormalities in screening assessments (e.g., ALT >1.5×ULN, creatinine >ULN, neutrophils <1.5×10⁹/L, platelets <100×10⁹/L, hemoglobin <100 g/L);
21. Pregnant/lactating women or positive pregnancy test;
22. Needle phobia, poor venous access, or intolerance to venipuncture;
23. Any other condition deemed by investigators to preclude compliance or safe participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
The occurrence of adverse events (AEs)/serious adverse events (SAEs) (including injection site reactions) from administration to the last visit | 105 days
  Types of Adverse Events / Serious Adverse Reactions
The occurrence of adverse events (AEs)/serious adverse events (SAEs) (including injection site reactions) from administration to the last visit | 105Days
  Incidence of Adverse Events/Serious Adverse Reactions
The occurrence of adverse events (AEs)/serious adverse events (SAEs) (including injection site reactions) from administration to the last visit | 105Days
  Severity of Adverse Events (AEs)/Serious Adverse Reactions (SARs)
The occurrence of adverse events (AEs)/serious adverse events (SAEs) (including injection site reactions) from administration to the last visit | 105Days
  Relationship of Adverse Events (AEs)/Serious Adverse Reactions (SARs) to the Investigational Product
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：P Wave
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：QRS Complex
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：T Wave
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：U Wave
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：PR Interval
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：QT Interval
The clinical significance of changes in observation indicators at different time points after drug injection compared to pre-administration. | 105Days
  12-lead electrocardiogram examination：ST Segment
Clinically significant changes in laboratory parameters from baseline at specified timepoints post-dosing | 105Days
  Complete Blood Count (CBC)

SECONDARY OUTCOMES:
Pharmacokinetic Endpoints | 105Days
  Cmax: Maximum plasma concentration
Pharmacokinetic Endpoints | 105Days
  AUC~0-t: Area under the curve from 0 to last measurable timepoint
Pharmacokinetic Endpoints | 105Days
  AUC~0-∞: Area under the curve extrapolated to infinity
Pharmacokinetic Endpoints | 105Days
  T~max: Time to reach Cmax
Pharmacokinetic Endpoints | 105Days
  t~1/2: Elimination half-life
Pharmacokinetic Endpoints | 105Days
  CL/F: Apparent clearance
Pharmacokinetic Endpoints | 105Days
  Vz/F：Apparent Volume of Distribution during Terminal Phase
Pharmacokinetic Endpoints | 105Days
  MRT：Mean Residence Time
Pharmacodynamic Endpoints | 0 to 12 hours
  Change in tetanus-neutralizing antibody titer from baseline within 12 hours post-dose across treatment groups
Pharmacodynamic Endpoints | 105Days
  Percentage of participants with anti-tetanus toxin neutralizing antibody titers ≥0.01 IU/mL and ≥0.1 IU/mL at each timepoint post-dose across treatment groups
Pharmacodynamic Endpoints | 105Days
  Percentage of participants with anti-tetanus toxin neutralizing antibody titer increases from baseline ≥0.01 IU/mL and ≥0.1 IU/mL at each timepoint post-dose across treatment groups
Exposure-Response Analysis, E-R Analysis | 105Days
  Exposure-response (E-R) analysis of serum drug concentrations versus anti-tetanus toxin neutralizing antibody titers at each post-dose timepoint across treatment groups
Immunogenicity Endpoints | 105Days
  Anti-drug antibody (ADA) titers against the investigational drug (recombinant human anti-tetanus toxin monoclonal antibody) in serum at each post-dose timepoint across treatment groups
Immunogenicity Endpoints | 105Days
  Incidence of anti-drug antibodies (ADA) against the investigational drug (recombinant human anti-tetanus toxin monoclonal antibody) in serum post-dose across treatment groups
Immunogenicity Endpoints | 105Days
  In participants who tested positive for anti-drug antibodies (ADA), the incidence of neutralizing antibodies (NAb) was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianchang He, Principal Investigator — Yunnan Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Lanzhou Institute of Biological Products Co., Ltd., Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided